CLINICAL TRIAL: NCT06852131
Title: Comparison of Surgical Treatment for Carpal Tunnel Syndrome with Corticosteroid Injection and Platelet-Rich Plasma Injection
Brief Title: Carpal Tunnel Syndrome Treatment: Surgery Vs. Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Yusuf Kıratlıoğlu, ankara university, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: İ02-82-22
Record Dates: First submitted 2025-02-18; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2022-01

CONDITIONS: Carpal Tunnel Syndrome (CTS)
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- surgery group (Active Comparator)
  Interventions: Procedure: open carpal tunnel surgery
- steroid injection group (Active Comparator)
  Interventions: Procedure: Steroid Injection
- prp injection group (Active Comparator)
  Interventions: Procedure: PRP injection

INTERVENTIONS:
Procedure: open carpal tunnel surgery — open carpal tunnel surgery
  Arms: surgery group
Procedure: Steroid Injection — triamsinolon injection
  Arms: steroid injection group
Procedure: PRP injection — PRP injection
  Arms: prp injection group

SUMMARY:
This prospective randomized controlled study included 68 patients (aged 18-70) with mild to moderate carpal tunnel syndrome (CTS), randomized into three groups: surgical treatment (25 patients, 25 wrists), corticosteroid (CS) treatment (20 patients, 32 wrists), and platelet-rich plasma (PRP) treatment (23 patients, 35 wrists). Diagnosis was confirmed through clinical evaluation and electrodiagnostic (EDX) testing, with assessments including the Visual Analog Scale (VAS), Boston Carpal Tunnel Questionnaire (BCTQ), ultrasonographic median nerve cross-sectional area (CSA) and flattening ratio (FR), and sensory/motor conduction parameters. Treatments were ultrasound-guided CS (1 mL triamcinolone, 40 mg/mL) or PRP (1 mL extracted from centrifuged venous blood) injections, while surgical treatment involved standard open carpal tunnel release using the WALANT (Wide Awake Local Anesthesia No Tourniquet) technique. Follow-ups were conducted at 1, 3, and 6 months, and the study was ethically approved with informed patient consent.

ELIGIBILITY:
Inclusion Criteria:

minimum of 3 months duration of symptoms and mild to moderate CTS

Exclusion Criteria:

* 1) Patients with severe CTS diagnosed with EMG or the presence of thenar atrophy, 2) Polyneuropathy, 3) Previous injection therapy for CTS, 4) Previous CTS surgery, 5) Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Electrophysiological studies | 1-3-6 months
  All EDX were performed using the Medtronic Key-Point EMG device (Denmark) by a neurology expert. Sensory and motor conduction studies of the median nerve and sensory conduction studies of the ulnar nerve were performed using standard techniques of supramaximal stimulation. Stimulation intensity was increased (3 mA for sensory or motor studies) each time until supramaximal stimulation was reached and maximal action potential was achieved. Sensory nerve conduction studies were performed with an antidromic method. Median nerve sensory nerve conduction velocity (SNCV) and sensory nerve action potential (SNAP) amplitude were calculated by recording from thumb and ulnar nerve from the 5th finger. Median nerve compound muscle action potential (CMAP) amplitude and distal motor latency (DML) were recorded from the abductor pollicis brevis Comparing with our clinical neurophysiology laboratory's normal values, the patients with only abnormal SNCVs (small or slow) with normal motor conduction we
ultrasonography | 1-3-6 months
  In both measurements and injections, the patients were positioned as follows: shoulder in a neutral position, elbow at 90º flexion, forearm supinated, wrist in slight extension, and fingers in semi-flexion. For examination, a linear array probe portable US device (Clarius, L7 HD3 Linear Scanner) was used. Median nerve CSA was measured using the manual trace method in axial view in the proximal carpal tunnel (at the scaphoid-pisiform level), where the median nerve's largest enlargement was found. The mean of cross-sectional area (CSA) was calculated using three consecutive measurements (mm²) and recorded. Flattening ratio (FR) was calculated by dividing the transverse diameter of the nerve by its anteroposterior diameter.
Boston carpal tunnel Questionnaire | 1-3-6 months
Visual Analog Scale | 1-3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No